CLINICAL TRIAL: NCT06652750
Title: Evaluating the Safety and Effectiveness of 5G Cloud Follow-up for Cardiovascular Implantable Electronic Devices: a Prospective, Paired, Self-controlled, Non-inferiority, Multicenter Clinical Trial
Brief Title: Evaluating the Safety and Effectiveness of 5G Cloud Follow-up for Cardiovascular Implantable Electronic Devices
Acronym: CIED-CARE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third People's Hospital of Chengdu (Other)
Responsible Party: Principal Investigator, Lin Cai, Professor of Department of Cardiology, The Third People's Hospital of Chengdu
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2024-S-182-01
Record Dates: First submitted 2024-10-10; First posted 2024-10-22 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: Sick Sinus Syndrome; Atrioventricular Block, Second and Third Degree; Heart Failure
Keywords: pacemaker; implantable cardioverter defibrillator; cardiac resynchronization therapy; follow up; remote programming; in-office follow-up
MeSH Terms: conditions — Sick Sinus Syndrome; Atrioventricular Block; Neoplasm Metastasis; Heart Failure

STUDY DESIGN:
Intervention Model Description: During each session, the CIED patient undergoes both the experimental and control methods.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 5G cloud follow-up & Routine follow-up (Experimental): CIED patients undergo both 5G cloud follow-up and routine in-office follow-up during each visit.
  Interventions: Other: Routine Management; Device: 5G Cloud Follow-up

INTERVENTIONS:
Other: Routine Management — Conducting routine in-office follow-up for CIED paitents
Device: 5G Cloud Follow-up — This study employed a 5G-cloud follow-up platform, a research tool that allows a device specialist to test, and program CIEDs in real-time from a remote location via an internet connection or mobile wireless network. Consistent with of the 5G remote support terminal externally connected to the programmer, a PAD was installed with a 5G-cloud follow-up app. The onsite medical staff began the cloud follow-up session by contacting the remote device specialist via video call. The connection to the CIED was made by the medical staff through the use of a standard programmer. He was in charge of turning on the programmer and applying the programmer wand to the patient's device. After an initial introduction, communication was established and continued via the wand connection. The remote device specialist logged into the 5G-cloud follow-up app with two-step verification. The remote device specialist then had complete control of the programmer to check and reprogram the device as needed.

SUMMARY:
Objective: This clinical study employs a prospective, paired, self-controlled, non-inferiority, multicenter research design to assess the safety and efficacy of utilizing 5G cloud follow-up for CIED in parameters monitoring and remote programming post-implantation.

Participants will:

undergo regular clinic follow-up visits in accordance with the guidelines undergo routine in-office follow-up and 5G cloud follow-up during each regular clinic visit

DETAILED DESCRIPTION:
Background: Cardiovascular implantable electronic devices (CIED) include pacemakers, implantable cardioverter defibrillators (ICD), cardiac resynchronization therapy (CRT) pacemakers and defibrillators, implantable cardiac event recorders (ICM), and implantable cardiovascular monitors. They are mainly used for the diagnosis, monitoring, and treatment of bradycardia, tachycardia, and heart failure (HF). There are currently two main methods of follow-up: routine in-office follow-up and remote monitoring (RM). Routine in-office follow-up is the most commonly used method in China, whereby professional doctors and/or manufacturer engineers conduct follow-ups under the guidance of physicians. Remote monitoring (RM) allows patients to be remotely monitored at home or elsewhere when a communication network is available, receiving periodic alerts related to the patient. Remote monitoring (RM) can provide timely and accurate CIED data and information, promptly alerting clinical doctors to any issues. However, a drawback is that patients still need to visit the hospital for device parameter adjustments, so it only partially fulfills the functions of routine in-office follow-up. Of note, in the past three years, some domestic clinical centers in China have begun exploring the application of 5G cloud follow-up remote programming (5G Cloud Follow Up) in various patient follow-up scenarios. With the comprehensive deployment of 5G networks in China, central hospitals with specialized device programmers can establish one-to-one or one-to-many regional collaborative cloud follow-up systems with primary hospitals lacking follow-up technician through 5G networks. CIED patients only need to visit nearby primary hospitals to complete regular device follow-ups. Currently, excellent research results have been obtained in the quality control of the CIED follow-ups of a single provincial medical consortium system mainly consisting of major implantation centers. However, there is still a lack of verification results for 5G cloud follow-up remote programming in a medical consortium (MC) model covering various administrative regions in China and different levels of primary hospitals. This study will compare the safety and effectiveness of using 5G cloud follow-up remote programming in different administrative regions and levels of primary hospitals in China with routine in-office follow-ups.

Objective:

This clinical study employs a prospective, paired, self-controlled, non-inferiority, multicenter research design to assess the safety and efficacy of utilizing 5G cloud follow-up for CIED in parameters monitoring and remote programming post-implantation.

Participants will:

undergo regular clinic follow-up visits in accordance with the guidelines undergo routine in-office follow-up and 5G cloud follow-up during each regular clinic visit

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years, gender unspecified;
2. Patients who have not undergone their first clinic follow-up after the implantation of cardiovascular implantable electronic devices (CIED); Note: In this study, CIED includes pacemakers, implantable cardioverter defibrillators (ICD), cardiac resynchronization therapy pacemakers (CRT-P) and defibrillators (CRT-D), excluding implantable cardiac event recorders (ICM) and implantable cardiovascular monitors.
3. Willing to participate in this clinical study and have signed the informed consent form in writing.

Exclusion Criteria:

* Exclusion Criteria:

If meeting any of the following, the individual cannot be included:

1. Life expectancy < 1 year.
2. Inability to cooperate with treatment or follow-up, such as having mental illness.
3. Participated in other clinical studies within 30 days before enrollment. Other situations that the researcher deems unsuitable for inclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 688 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Parameter Measurement Consistency | through study completion, an average of 1 year
  Subjects underwent in-office follow-up and 5G cloud follow-up to test battery parameters (battery voltage, battery current, and magnet frequency) and lead parameters (amplitude, pacing threshold, and impedance) in the immediate postoperative period, prior to discharge from the hospital, and within 1 month of implantation, within 1 to 3 months of implantation, at 6 months of implantation, and at 12 months of implantation, respectively. The consistency of each parameter measured at both follow-up modalities was analyzed at the end of the trial by regression fitting equations and Pearson correlation coefficients.

SECONDARY OUTCOMES:
Parameter Measurement Time | through study completion, an average of 1 year
  During each follow-up, all subjects undergo separate routine in-office follow-ups and 5G cloud follow-ups. The time taken from the beginning of device interrogation to the completion of parameter testing is recorded for each follow-up.
Program Completion Rate | through study completion, an average of 1 year
  Evaluation Approach: Participants undergo both in-person clinic follow-up and 5G cloud follow-up during each appointment. Researchers will evaluate and programe the device in accordance with the current guidelines. The assessment of program completion will be conducted through the Program Control Completion Assessment Form.
  Completion Criteria: If all parameter reprogramming statuses are indicated as "Yes", the program control session will be deemed as complete. In cases where any program control completion status is marked as "No", the session's program control will be considered incomplete.
  Program Completion Rate is calculated as follows: the number of successful programming / the total number of programming
adverse events | through study completion, an average of 1 year
  Subjects are observed and recorded at any time during the study process after enrollment. Summarize the occurrence of adverse events and calculate the rate of adverse events. Participants will be continuously monitored and documented during each follow-up session. The adverse event is defined according to the "Guidelines for Reporting Adverse Events and Device Defects" in the present study. Investigators will record and summarize the occurrence of adverse events and determine the rate of adverse event incidence. The rate of adverse event is calculated as the number of participants occurring adverse event/ the total number of the participants.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Sun Yat-sen Memorial Hospital, Guangzhou, Guangdong
  - The Third People's Hospital of Chengdu, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: Undecided
The datasets in the study might be available upon reasonable request.

REFERENCES:
- [Background] Xiong S, Qin S, Tong L, Long Y, Luo Y, Feng Q, Peng X, Jiang M, Xiong F, Li J, Zhang Y, Zhang Z, Liu H, Cai L. The clinical use of remote parameter testing during cardiac implantable electronic devices implantation procedures: a single center, randomized, open-label, non-inferiority trial. Front Cardiovasc Med. 2024 Mar 22;11:1364940. doi: 10.3389/fcvm.2024.1364940. eCollection 2024. PMID 38586175
- [Background] Xiong S, Li J, Tong L, Hou J, Yang S, Qi L, Chen X, Luo Y, Zhang Z, Liu H, Cai L. Realtime Remote Programming in Patients Carrying Cardiac Implantable Electronic Devices Requiring Emergent Reprogramming. Front Cardiovasc Med. 2022 May 16;9:871425. doi: 10.3389/fcvm.2022.871425. eCollection 2022. PMID 35651905
- [Background] Tong L, Xiong S, Hou J, Li J, Qin S, Zhang Y, Yang S, Qi L, Chen X, Luo Y, Zhang Z, Deng H, Liu H, Cai L. Cloud Follow-Up in Patients With Cardiovascular Implantable Electronic Devices: A Single-Region Study in China. Front Cardiovasc Med. 2022 May 9;9:864398. doi: 10.3389/fcvm.2022.864398. eCollection 2022. PMID 35615564
- [Background] Tong L, Long Y, Xiong S, Li J, Huang W, Liu H, Cai L. Application of Postoperative Remote Follow-Up of CIED Based on the 5G Cloud Technology Support Platform in Areas With Underdeveloped Medical Resources. Front Cardiovasc Med. 2022 Jun 17;9:894345. doi: 10.3389/fcvm.2022.894345. eCollection 2022. PMID 35783847